CLINICAL TRIAL: NCT02555150
Title: A Randomized, Phase 3, Double-Blind, Crossover Comparison of PRC-063 and Lisdexamfetamine in the Driving Performance of Adults With ADHD
Brief Title: A Comparison of PRC-063 and Lisdexamfetamine in the Driving Performance of Adults With ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rhodes Pharmaceuticals, L.P. (Industry)
Collaborators: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 063-013
Record Dates: First submitted 2015-08-28; First posted 2015-09-21 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PRC-063 (Active Comparator): Titration during which subjects will be titrated from a starting dose of 45 mg/day (dosed once daily) of PRC-063 oral capsules up to his/her final dose (45, 70 or 100 mg/day of PRC-063). This phase will be 10 to 21 days long.
  Interventions: Drug: PRC-063; Drug: Placebo
- lisdexamfetamine dimesylate (Active Comparator): Titration during which subjects will be titrated from a starting dose of 30 mg/day of lisdexamfetamine up to his/her final dose (30, 50 or 70 mg/day of LDX). This phase will be 10 to 21 days long.
  Interventions: Drug: lisdexamfetamine dimesylate; Drug: Placebo
- Placebo (Placebo Comparator): Subjects will be dosed once daily with a placebo oral capsule for 10 to 21 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PRC-063 — Oral extended-release capsule
  Arms: PRC-063
Drug: lisdexamfetamine dimesylate — Oral capsule
  Arms: lisdexamfetamine dimesylate
Drug: Placebo — Oral placebo capsule

SUMMARY:
The purpose of this randomized, double-blind, crossover study is to compare two long-acting stimulant formulations-once-daily PRC-063 and once-daily lisdexamfetamine (LDX)-through a 15-hour period on driving performance, as measured with a driving simulator, in adult patients with ADHD.

DETAILED DESCRIPTION:
Young adult drivers with Attention Deficit Hyperactivity Disorder (ADHD) will be compared on a driving simulator after taking PRC-063 or LDX in a repeated-measure, randomized, doubleblind, crossover study design. Each subject will be randomized to receive up to a 21-day course of PRC-063 followed by up to a 21 day course of LDX or vice versa. There will be no washout between treatments. On days 1 through 7, subjects will receive the lowest dose (45 mg of PRC-063 or 30 mg of LDX) of study medication. On days 8 through 14, subjects will receive the middle dose (70 mg of PRC-063 or 50 mg of LDX). On days 15 through 21, subjects will receive the highest dose (100 mg of PRC-063 or 70 mg of LDX). During Days 1 through 21, if a subject is responding satisfactorily to medication, he or she may remain on that daily dose. Driving laboratory testing will be conducted between Day 17 and Day 21. Following the laboratory testing, the subject will begin a second titration of the alternate treatment, starting on Day 22 through Day 28 at the lowest dose (45 mg of PRC-063 or 30 mg of LDX) of study medication, Day 29 through Day 35 on the middle dose (70 mg of PRC-063 or 50 mg of LDX) and Day 36 through Day 42 on the highest dose (100 mg of PRC-063 or 70 mg of LDX). During Days 22 through 42, if a subject is responding satisfactorily to medication, he or she may remain on that daily dose. Following titration with the second treatment, subjects will attend a second driving laboratory testing, conducted between Day 38 to Day 42. Subjects will subsequently attend a safety and study termination visit.

ELIGIBILITY:
Inclusion Criteria:

Male or non-pregnant, non-nursing female at least 18 years of age and less than or equal to 25 years of age with a valid driver's license and at least six months of driving experience with driving activity at least twice per week.

ADHD diagnosis, inattentive, hyperactive/impulsive or combined, as defined by the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) based on clinician assessment using the Structured Clinical Interview for DSM Disorders (SCID).

Dissatisfaction with his or her current pharmacological therapy for treatment of ADHD or not currently receiving pharmacological therapy for ADHD. Inclusion of subjects naïve to pharmacological therapy for ADHD is permitted.

Exclusion Criteria:

Known to be non-responsive to methylphenidate or lisdexamfetamine treatment. Nonresponse is defined as methylphenidate or lisdexamfetamine use at various doses for a phase of at least four weeks at each dose with little or no clinical benefit in the last 10 years.

Having a history of motion, sea or big screen (e.g. IMAX) sickness, in order to avoid possible Simulation Adaptation Syndrome.

Subject has a known family history of sudden cardiac death or ventricular arrhythmia.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Tactical Driving Quotient (TDQ) | At 21 days (Visit 9)
  The primary outcome measure will be the Tactical Driving Quotient (TDQ) between treatments.
  The TDQ is an accumulative effect size across multiple driving variables collected during the driving simulation, including: summed standard deviations of steering, driving off the road, veering across the midline, inappropriate braking while on the open road, missed stop signs, exceeding speed limit, standard deviation of speed, time at stop sign deciding when to turn left and time to complete left turns. A higher TDQ score reflects better driving skill. A TDQ of 100 represents average driving and the standard deviation of normal distribution is 15. The normal range of driving (+/- 1.0 SD) is 85 to 115. A TDQ of less than 100 represents worse than average driving (e.g., a TDQ of 115 represents driving performance 1 SD better than average) and a TDQ of greater than 100 represents better than average driving.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | Participants will be followed for the duration of the study, an expected average of 10 weeks
  Summary of adverse events reported during the study
Columbia Suicide Severity Rating Scale (CSSRS) | At one week and nine weeks of the study
  A Columbia Suicide Severity Rating Scale (CSSRS) assessment will be administered by the investigator to all study participants

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Reiz, Study Director — Purdue Pharma LP
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No